CLINICAL TRIAL: NCT01993589
Title: Effect of Paracetamol, Dexketoprofen Trometamol, Lidocaine Spray, Pethidine and Diclofenac Sodium Application for Pain Relief During Fractional Curettage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Açmaz, MD, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: {kayseriERH}
Record Dates: First submitted 2013-11-09; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Pain and Curettage
Keywords: Curettage; analgesia; paracetamol; lidocaine; Dexketoprofen trometamol; pethidine; diclofenac.
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control group (No Intervention): Control group
- Pain reliever (Active Comparator): 1000 mg paracetamol (Parol 1 g Atabay ilaç Turkey)
  Interventions: Drug: comparison of pain relievers during curattage
- Dexketoprofen trometamol (Active Comparator): 25 mg oral Dexofen Atabay ilaç Turkey
  Interventions: Drug: comparison of pain relievers
- Lidocaine spray (Active Comparator): 2 puff on cervical mucosa (Xylocain Pump 100 Mg 50 Ml Sprey Astra Zeneca)
  Interventions: Drug: comparison of pain relievers during curattage
- pethidine (Active Comparator): Aldolan 100 mg Liba Laboratuarı İstanbul Turkey
  Interventions: Drug: comparison of pain relievers during curattage
- diclofenac sodium (Active Comparator): Dicloron amp 75 mg Deva İlaç Levent İstanbul/Turkey
  Interventions: Drug: comparison of pain relievers during curattage

INTERVENTIONS:
Drug: comparison of pain relievers during curattage
  Arms: Pain reliever
Drug: comparison of pain relievers
  Arms: Dexketoprofen trometamol
Drug: comparison of pain relievers during curattage
  Arms: Lidocaine spray
Drug: comparison of pain relievers during curattage
  Arms: pethidine
Drug: comparison of pain relievers during curattage
  Arms: diclofenac sodium

SUMMARY:
Patients frequently experience pain from moderate to severe during gynecologic procedures. This study is a prospective, randomized, placebo-controlled trial and aimed to investigate the analgesic efficacy of preoperative oral dexketoprofen trometamol, intravenous paracetamol, lidocaine spray, pethidine and diclofenac sodium on fractional curettage procedure.

DETAILED DESCRIPTION:
A total of 144 mutiparous subjects randomly allocated one of six groups. The first group (control group) consisted of 22 participants and they did not receive any treatment. The second group consisted of 26 participants receiving oral 25 mg dexketoprofen trometamol. The third group consisted of 23 participants receiving 2 puff lidocaine sprays on cervical mucosa. The forth group consisted of 25 participants receiving 100 mg pethidine. The fifth group consisted of 23 participants receiving 1000 mg intravenous paracetamol and the sixth group consisted of 25 participants receiving diclofenac sodium.

ELIGIBILITY:
Inclusion Criteria:

* multiparous participants
* abnormal uterine bleeding
* postmenopausal bleeding
* myoma uteri causing menometrorrhagia
* cervical polyp
* tamoxifen treatment for breast cancer
* adnexial mass

Exclusion Criteria:

* abortions
* pregnancy
* primiparity
* diabetes mellitus
* tendency to bleed such as thrombocytopenia
* factor deficiency
* functional disorders of platelets

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Education and Research Hospital of Medicine, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Acmaz G, Bayraktar E, Aksoy H, Baser M, Yilmaz MO, Muderris II. Effect of paracetamol, dexketoprofen trometamol, lidocaine spray, pethidine & diclofenac sodium application for pain relief during fractional curettage: A randomized controlled trial. Indian J Med Res. 2015 Oct;142(4):399-404. doi: 10.4103/0971-5916.169197. PMID 26609031